CLINICAL TRIAL: NCT00510822
Title: Safety and Efficacy of Cimicoxib, a Selective COX-2 Inhibitor, in Combination With Sertraline Compared to Sertraline Combined With Placebo in Treatment of Major Depression
Brief Title: Cimicoxib for the Treatment of Major Depression (SECIM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affectis Pharmaceuticals AG (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFX-01; EudraCT-No. 2007-001335-54
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Major Depression
Keywords: Cimicoxib; Cox-2 inhibitor; Sertraline
MeSH Terms: conditions — Depressive Disorder, Major | interventions — cimicoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo + Sertraline
  Interventions: Drug: Placebo
- Cimicoxib (Experimental): Sertraline + Cimicoxib
  Interventions: Drug: Cimicoxib

INTERVENTIONS:
Drug: Cimicoxib — 50 mg per tablet, bid (total daily dose 100 mg)
  Other Names: AFX
  Arms: Cimicoxib
Drug: Placebo — tablet
  Other Names: PLC
  Arms: Placebo

SUMMARY:
This multicenter study aims to investigate the safety and efficacy of cimicoxib, a selective COX-2 inhibitor, in combination with sertraline compared to sertraline combined with placebo in patients with major depression. This clinical study is based on the assumption that adjunctive treatment of major depression with a COX-2 inhibitor may be beneficial.

DETAILED DESCRIPTION:
Adult patients of both gender, aged between 18 and 60 years diagnosed with major depression by a psychiatrist and a HamD-17 score ≥ 22 will be enrolled. All patients will undergo a wash out period of 3 days (without e.g. medication or antidepressant medication) prior to receiving sertraline combined with cimicoxib or placebo. In the exceptional case where in opinion of the investigator concomitant psychotic treatment is needed, up to 3 mg lorazepam daily can additionally be administrated during this period and the first two weeks of treatment.Assessment of HamD-17 will be performed by trained psychiatric raters before wash out and at week 0 (baseline) prior to the treatment. If the HamD-17 score decreases to less than 22 at the second rating patients will be excluded from study.Patient must be in-patients during the wash out period and the first two weeks of treatment. Upon recommendation of the investigator, participants can become out-patients with ambulatory care at day clinics after the first two weeks of treatment.At baseline (week 0) patients will be randomised to one of the following treatment arms:· 50 mg of sertraline (one tablet/unblinded) daily plus cimicoxib (one tablet-50mg) twice daily.· 50 mg of sertraline (one tablet/unblinded) daily plus placebo (one tablet) twice daily If at study visit 3 (i.e. after 3 weeks of treatment) the baseline therapy dose of 50 mg of sertraline daily is considered as not therapeutically sufficient (increase of HamD-17 by more than 20% compared to baseline), it can be increased to 100 mg daily at the discretion of the investigator. The decision by the investigator to increase sertraline dose to 100 mg daily is allowed only at study visit 3 and is not permitted at any other time during the study.During the double-blind period, study visits will take place every week until week 6 and clinical psychiatric and safety assessments will be performed. Four weeks after the end of treatment the investigators or their designees will call the patients to capture information on how the patients feel and to assess if the patients experienced any SAE/AEs (e.g. hospitalisations).

ELIGIBILITY:
Inclusion Criteria:

* Major depression diagnosed by psychiatrist
* DSM IV TR: 296.2x single depressive episode or 296.3x recurrent depressive episode
* HamD-17 score ≥ 22

Exclusion Criteria:

* Psychotic depression, bipolar disorder, obsessive compulsive disorder, anxiety disorder, personality disorder, drug or alcohol abuse, schizoaffective disorders, schizophrenia
* All DSM IV TR Axis-I disorders except depression
* All DSM IV TR Axis-II disorders without exception
* Unsuccessful treatment with more than 2 antidepressant medications
* Concomitant use of psychotropic drugs, including mood stabilizers
* Immediate risk of suicidal behaviour
* Women who are pregnant, breast feeding or planning to become pregnant during the course of study, Women who are not post-menopausal, surgically sterilized or using an effective method of contraception
* Any history of cardiovascular disease (e.g. angina, heart attack, stroke, congestive heart failure), uncontrolled high blood pressure, documented peripheral arterial insufficiency and symptomatic, clinically significant claudication, or a history of peripheral arterial embolism
* History of coronary heart disease (CHD) or any other heart disease
* History of upper or lower gastrointestinal (GI) ulceration, perforation and/or obstruction
* History of upper or lower GI bleeding within the previous year
* History of inflammatory bowel disease

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 169 (Actual)
Dates: Start 2007-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
• Mean change on the total score of the Hamilton Depression Rating Scale (HamD-17) from baseline to endpoint (Week 6). | 6 Weeks

SECONDARY OUTCOMES:
• Changes from baseline to interim weekly visits (week 1 to 5) in HamD-17 score • Clinical Global Impression (CGI) score • Montgomery Asberg Depression Rating Scale (MADRS) score • Response rate, remission rate and drop out rate. • Onset of | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Rüdiger, Study Director — Affectis Pharmaceuticals AG
Locations (25):
- Austria (2):
  - Landeskrankenhaus Klagenfurt, Abteilung für Psychiatrie und Psychotherapie, Klagenfurt
  - Gemeinnützige Salzburger Landeskliniken Betriebsgesellschaft mbH, Salzburg
- Czechia (6):
  - Faculty Hospital Brno, Brno
  - Hospital Ceske Budejovice, České Budějovice
  - Pardubice Regional Hospital, Pardubice
  - 1st Medical Faculty Prague, Prague
  - Prague Psychiatric Centrum, Prague
  - Masaryk Hospital, Ústí nad Labem
- Germany (17):
  - Charite - Center for Psychiatry and Psychotherapy, Berlin
  - LWL-Universitätsklinik Bochum, Bochum
  - University Bonn, Center for Psychiatry and Psychotherapy, Bonn
  - Klinik für Psychiatrie und Psychotherapie der Universität zu Köln, Cologne
  - Carl Gustav Carus University Dresden, Center for Psychiatry and Psychotherapy, Dresden
  - Georg-August-University Goettingen, Department of Psychiatry and Psychotherapy, Göttingen
  - Hospital Guenzburg, Center for Psychosomatic Medicine, Günzburg
  - University Jena, Center for Psychiatry and Psychotherapy, Jena
  - Fachklinik Katzenelnbogen, Limburg An Der Lahn (Katzenelnbogen)
  - Otto-von-Guericke University Magdeburg, Department of Psychiatry, Psychotherapy and Psychosomatic Medicine, Magdeburg
  - Klinikum der Johannes Gutenberg-Universität Mainz, Mainz
  - Zentralinstitut für Seelische Gesundheit, Klinik für Psychiatrie und Psychotherapie, Mannheim
  - Ludwig-Maximilians University Munich, Munich
  - Max Planck Institute of Psychiatry, Munich
  - Center for Psychiatry and Psychotherapy, University of Muenster, Münster
  - Bezirksklinikum Regensburg, Regensburg
  - Ernst Moritz Arndt University of Greifswald, Center for Psychiatry and Psychotherapy, Stralsund